CLINICAL TRIAL: NCT00598767
Title: Multimodality 3D Imaging and Wireless Technologies To Enhance Medical Care in Space
Brief Title: Three Dimensional Imaging and Wireless Technologies to Enhance Medical Care in Space
Status: Terminated | Type: Observational
Why Stopped: funding issues
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NSBRI NCC9-59-172 #2
Record Dates: First submitted 2007-12-26; First posted 2008-01-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-01

CONDITIONS: Aortic Valve Insufficiency; Aortic Stenosis
Keywords: Aortic valve insufficiency; Aortic valve stenosis; 3D echocardiogram; 3D computed tomography
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
NASA has outlined the most urgent threats to life and health in manned spaceflight. One of the threats is the risk of trauma and acute medical problems. One of the most important provisions of acute and chronic medical services in space is the availability of high quality diagnostic imaging with the potential for either ground based or onsite interpretation. The principle diagnostic imaging modality for space crew use in space will be ultrasound. The aim of the study is as follows:

-To use state of the art 3 dimensional CT scanner to acquire images for segmentation and registration supplying a template to judge physiologic or pathologic changes observed in space with 3D ultrasound

DETAILED DESCRIPTION:
In its Bioastronautics Critical Path Roadmap Baseline Document, NASA has outlined the most urgent threats to life and health in manned spaceflight currently in need of countermeasures development. This proposal specifically addresses one of four critical risks directly, that being the risk of trauma and acute medical problems, ID# 43 in the Clinical Capabilities discipline area. Critical for the provision of acute and chronic medical services in space is the availability of high quality diagnostic imaging, with either ground-based or autonomous interpretation. While development of novel sensor technology is actively pursued within the NSBRI, it is clear that for the foreseeable future, the principal diagnostic imaging modality for crew use in space will be ultrasound. For the past six years, the Cleveland Clinic has worked with NASA and NSBRI in a comprehensive program to develop ultrasonographic capabilities for use in manned space flight. Recent work has focused on enhancement of these capabilities, including 3D imaging and novel compression and registration techniques for assessing change over time in ultrasonic images. We now propose to extend these capabilities in very significant ways, capitalizing on dramatic recent advances in telecommunications and computerization to better address the critical countermeasures identified. Among the convergent trends in ultrasound that we seek to capitalize on are the following: most commonly applied diagnostic imaging test; Miniaturization; file storage; telemedicine; wireless telemetry; therapeutic use; real-time 3D.

We propose to extend our work with the following Specific Aims:

1. Extension of our longstanding research in 3D ultrasound with a recently developed third generation machine small enough to fit on the ISS, allowing more comprehensive imaging to be done with less operator expertise.
2. Utilization of a ultrafast 3D CT scanner to acquire full body 3D images for segmentation and registration with subsequently acquired 3D ultrasound images, modelling future missions for ground-based 3D CT or MRI could provide a template to judge physiologic or pathologic changes observed in space with 3D ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Aortic regurgitation or aortic stenosis and scheduled for repair or replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Cleveland Clinic undergoing aortic valve repair or replacement
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2003-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To use and compare state-of-the-art 3D CT scanner to acquire 3D images for segmentation and registration with subsequent acquired 3D ultrasound images | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jim D Thomas, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No